CLINICAL TRIAL: NCT04834596
Title: Detection and Automatic Segmentation of Liver Nodules in Patients With Colorectal
Brief Title: Detection and Automatic Segmentation of Liver Nodules in Patients With Colorectal Adenocarcinoma
Acronym: OOPS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021 OOPS
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Detection of Liver Metastases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients without hepatic metastases: hepatic scanner of 100 patients with colorectal cancer without hepatic metastases will be analysed
  Interventions: Other: retrospectives analysis on hepatic scanner
- patients with synchronous hepatic metastases: hepatic scanner of 100 patients with colorectal cancer with synchronous hepatic metastases will be analysed
  Interventions: Other: retrospectives analysis on hepatic scanner
- patients with metachronous hepatic metastases: hepatic scanner of 100 patients with colorectal cancer with metachronous hepatic metastases will be analysed
  Interventions: Other: retrospectives analysis on hepatic scanner

INTERVENTIONS:
Other: retrospectives analysis on hepatic scanner — hepatic scanner will be analysed by two radiologist and by the software

SUMMARY:
Evaluation of the diagnostic performance of artificial intelligence-based software for the detection of liver nodules on scanner in patients at risk of liver metastases of colorectal cancer

DETAILED DESCRIPTION:
The aim of this study is to evaluate the performance of a software for liver nodule detection in patients with colorectal cancer compared to the consensus of two radiologists analysis.

300 hepatic scanners will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients consecutively treated for colorectal cancer a
* Availability of imaging by injected abdominal scanner including at least one portal phase
* Age over 18

Exclusion Criteria:

* Patients with treatment of the hepatic nodule by ablation or previous hepatic surgery
* Imaging follow-up <12 months
* Non-interpretable scanner (artefact, injection quality, etc.)
* Patients with more than 10 liver metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-02 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-05-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the performance of the software for detection of hepatic nodules on CT scan of patients with colorectal cancer compared to a reference constituted by the evaluation established by two radiologists in consensus. | 1 month
  Number of nodules detected by the software compared to the reference method

CONTACTS AND LOCATIONS:
Locations (1):
- UHAngers, Angers, France

IPD SHARING:
Plan to Share IPD: No